CLINICAL TRIAL: NCT01737814
Title: Evaluation of Purified Poloxamer 188 in Vaso-Occlusive Crisis of Sickle Cell Disease (EPIC): A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Trial of MST-188 (Purified Poloxamer 188) Injection in Subjects With Sickle Cell Disease Experiencing Vaso Occlusive Crisis
Brief Title: Evaluation of Purified Poloxamer 188 in Vaso-Occlusive Crisis of Sickle Cell Disease (EPIC)
Acronym: EPIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mast Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MST-188-01
Record Dates: First submitted 2012-11-27; First posted 2012-11-30 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Vaso-occlusive Crisis; Sickle Cell Disease
Keywords: sickle cell disease; vaso-occlusive crisis
MeSH Terms: conditions — Vaso-Occlusive Crises; Anemia, Sickle Cell | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MST-188 (Experimental): MST-188 injection administered as a continuous infusion 100 mg/kg for 1 hour followed by 30 mg/kg/hr for up to 48 hours.
  Interventions: Drug: MST-188
- Saline (Placebo Comparator): Saline administered as a continuous infusion for up to 49 hours
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline
  Arms: Saline
Drug: MST-188
  Other Names: vepoloxamer
  Arms: MST-188

SUMMARY:
The purpose of this study is to evaluate whether MST-188 can reduce the duration of vaso-occlusive crisis (VOC) in subjects with sickle cell disease. The study will also evaluate whether MST-188 can reduce the frequency of rehospitalization of subjects due to a recurrence of VOC. Additionally, this study will compare the development of acute chest syndrome during VOC in subjects who receive MST-188 to those who do not receive MST-188.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 through 65 years
* Subject has a confirmed diagnosis of HbSS, HbSC, HbSβ+thal, or HbSβ0thal
* Subject is experiencing acute pain typical of vaso-occlusive crisis requiring treatment with parenteral analgesia
* Subject requires hospitalization

Exclusion Criteria:

* Subject has acute chest syndrome
* Subject's laboratory results indicate inadequate organ function
* Subject is pregnant or nursing an infant
* Subject had a painful crisis requiring hospitalization within the preceding 14 days or has experienced > 5 hospitalizations for VOC in the prior 6 months
* Subject has been transfused within the past 14 days
* Subject is hospitalized for a condition other than VOC
* Subject has complications related to SCD

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2013-05; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Reduction of the duration of vaso occlusive crisis (VOC) in subjects with sickle cell disease. | Study participants will be followed for the duration of hospital stay, an expected average of 4 days

SECONDARY OUTCOMES:
Re-hospitalization rate for VOC | Hospital discharge to 14 days post-discharge
Occurence of acute chest syndrome | Randomization to 120 hours after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Edwin L. Parsley, D.O., Study Director — Mast Therapeutics, Inc.
Locations (71):
- United States (50):
  - University of South Alabama, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - UCSF Benioff Children's Hospital, Oakland, California
  - University of California Davis Health System, Sacramento, California
  - Rady Children's Hosptial, San Diego, California
  - Harbor-UCLA Medical Center, Torrence, California
  - Al DuPont Hospital for Children, Wilmington, Delaware
  - Howard University, Washington D.C., District of Columbia
  - Children's Hospital of SouthWest Florida, Fort Myers, Florida
  - Joe Dimaggio Children's Hospital, Hollywood, Florida
  - University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital at the University of Illinois, Chicago, Illinois
  - Fort Wayne Lutheran Hospital, Fort Wayne, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa-Children's Hospital, Iowa City, Iowa
  - University of Louisville/Kosair Children's Hospital, Louisville, Kentucky
  - Our Lady of the Lake Children's Hospital, Baton Rouge, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - The Herman and Walter Samuelson Children's Hospital at Sinai, Baltimore, Maryland
  - Children's Hospital of Michigan-Wayne State University, Detroit, Michigan
  - Hurley Research Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Rutger's University, New Brunswick, New Jersey
  - NY Methodist, Brooklyn, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Golisano Children's Hospital at URMC, Rochester, New York
  - Bronx Lebanon Hospital, The Bronx, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Randall Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Medical University of South Carolina, Charleston, South Carolina
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - Cook's Children Hospital, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Virginia Medical Center, Charlottsville, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Hospital of Richmond, Richmond, Virginia
- Belgium (5):
  - Reearch Center, Antwerp
  - Research Center, Brussels
  - Research Center, Edgem
  - Research Center, Liège
  - Research Center, Montegnée
- Brazil (2):
  - Resaerch Center, Rio de Janerio
  - Research Center, São Paulo
- Research Center, Santo Domingo, Dominican Republic
- Research Center, Kingston, Jamaica
- Research Center, Irbid, Jordan
- Lebanon (2):
  - Research Center, Beirut
  - Research Center, Tripoli
- Oman (2):
  - Research Center - Child Health Department, Muscat
  - Research Center, Muscat
- Panama (3):
  - Research Center Hospital del Nino, Panama City
  - Research Center Hospital of Pediatric Specialities, Panama City
  - Research Center Metropolitan Hospital, Panama City
- Research Center, Madrid, Spain
- Turkey (Türkiye) (3):
  - Research Center, Adana
  - Research Center, Istanbul
  - Research Center, Mersin

REFERENCES:
- [Derived] Casella JF, Barton BA, Kanter J, Black LV, Majumdar S, Inati A, Wali Y, Drachtman RA, Abboud MR, Kilinc Y, Fuh BR, Al-Khabori MK, Takemoto CM, Salman E, Sarnaik SA, Shah N, Morris CR, Keates-Baleeiro J, Raj A, Alvarez OA, Hsu LL, Thompson AA, Sisler IY, Pace BS, Noronha SA, Lasky JL 3rd, de Julian EC, Godder K, Thornburg CD, Kamberos NL, Nuss R, Marsh AM, Owen WC, Schaefer A, Tebbi CK, Chantrain CF, Cohen DE, Karakas Z, Piccone CM, George A, Fixler JM, Singleton TC, Moulton T, Quinn CT, de Castro Lobo CL, Almomen AM, Goyal-Khemka M, Maes P, Emanuele M, Gorney RT, Padgett CS, Parsley E, Kronsberg SS, Kato GJ, Gladwin MT. Effect of Poloxamer 188 vs Placebo on Painful Vaso-Occlusive Episodes in Children and Adults With Sickle Cell Disease: A Randomized Clinical Trial. JAMA. 2021 Apr 20;325(15):1513-1523. doi: 10.1001/jama.2021.3414. PMID 33877274